CLINICAL TRIAL: NCT01188915
Title: Personalised Program for Women Treated for Hodgkin Disease : Risk Evaluation of Breast Cancer and Intensive Screening Program for Women at High Risk of Breast Cancer. PROPER/IPC 2010-001
Brief Title: Personalised Program for Women Treated for Hodgkin Disease
Acronym: PROPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PROPER/IPC 2010-001
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Hodgkin Disease; Breast Cancer
Keywords: Hodgkin disease; Breast cancer
MeSH Terms: conditions — Hodgkin Disease; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intensive screening (Experimental): annual breast cancer detection based on mammography, echography and RMI.
  Interventions: Procedure: intensive screening

INTERVENTIONS:
Procedure: intensive screening — Each year, women will have breast cancer detection based on mammography, echography and RMI. Questionaries will also be completed.

SUMMARY:
After treatment for Hodgkin disease, secondary cancer, in particular breast cancer induced by treatment, are the first cause of death.

The investigators will estimate the risk to develop breast cancer in this population of women treated for hodgkin disease, and will propose women at high rish to participate in an intensive screening program based on an annual detection based on mammography, echography, and RMI.

ELIGIBILITY:
Inclusion Criteria:

* women > 18 years
* treated for Hodgkin disease
* signed informed consent
* high risk of breast cancer

Exclusion Criteria:

* patients unable to have a regular follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-07; Primary Completion 2016-09 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
efficacy of the screening | 15 years
  The efficacy of the screening will be evaluated by the rate of early stage breast cancer detected. The rate of in situ, < 10 mm(T1b), and N0 will be estimated.

SECONDARY OUTCOMES:
interest | 1 month
  The rate of interest is the % of women at high risk who will accept the intensive screening
adhesion | 1 month
  The adhesion rate is the % of women who will effectively undergo the first screnning among the women who had accepted their participation in this intensive screening
compliance | 15 years
  The compliance will be evaluated yearly. The number of exam realised compared to the theoric number and the time between 2 exams will be estimated.
psychologic impact | 15 years
  The psychologic impact will be assessed yearly by questionnaries evaluating quality of life, anxiety and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: François EISINGER, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- François EISINGER, PhD, Marseille, France

REFERENCES:
- See also: institut Paoli-Calmettes web site — http://www.institutpaolicalmettes.fr/